CLINICAL TRIAL: NCT05655585
Title: Comparison of Mulligan Bent Leg Raise vs Active Release Technique in Patients With Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC -01393 Roheena Mustansar
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hamstring Injury
Keywords: pain; active release technique; mulligan bent leg raise; hamstring tightness
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Technique (Experimental): Participant will be in prone position on a couch with the therapist standing next to the patient. The patient is asked to flex the knee to 90 degree of the involved side. The therapist then applies gentle tension longitudinally to the hamstring muscle along the entire length while the patient actively moves his knee from flexion to extension
  Interventions: Other: Active Release Technique; Other: Mulligan Bent Leg Raise
- Mulligan Bent Leg Raise (Experimental): Participant was in supine lying on a high couch with the therapist in standing position lateral to the leg, which is to be stretched. Hip and Knee of the side to be stretched was bent at 90- 90 degree. Investigator places participant's flexed knee over his shoulder such that the popliteal fossa of the knee rest on his shoulder. A distraction (longitudinal traction force along the long axis of femur) was applied at the lower end of femur
  Interventions: Other: Active Release Technique; Other: Mulligan Bent Leg Raise

INTERVENTIONS:
Other: Active Release Technique — Participant will be in prone position on a couch with the therapist standing next to the patient. The patient is asked to flex the knee to 90 degree of the involved side. The therapist then applies gentle tension longitudinally to the hamstring muscle along the entire length while the patient actively moves his knee from flexion to extension
Other: Mulligan Bent Leg Raise — Participant was in supine lying on a high couch with the therapist in standing position lateral to the leg, which is to be stretched. Hip and Knee of the side to be stretched was bent at 90- 90 degree. Investigator places participant's flexed knee over his shoulder such that the popliteal fossa of the knee rest on his shoulder. A distraction (longitudinal traction force along the long axis of femur) was applied at the lower end of femur

SUMMARY:
The sedentary lifestyle of today's world, prolonged time period of sitting during office hours and educational setups do have an effect on the flexibility of bi-articular muscles. Hamstring flexibility is a significant variable as decreased extensibility has been suggested as a prejudicing feature for injuries, poor posture and non-specific low back pain.Active Release Technique (ART) is a soft tissue method that focuses on relieving tissue tension via the removal of fibrosis/adhesions which can develop in tissues as a result of overload due to repetitive use. These disorders may lead to muscular weakness, numbness, aching, tingling and burning sensations. ART has been reported to be both a diagnostic and a treatment technique.Mulligan's bent leg raise (BLR) is a stretching technique which is a modern progression in the treatment of hamstring tightness. It is indicated in hamstring tightness patients with backache having restricted or painful straight leg raise (SLR), leg pain above knee and it is very beneficial in the patients having gross bilateral limitations of straight leg raise. It stretches the lower extremity muscles in combination of hamstring, adductors and rotators

DETAILED DESCRIPTION:
The hamstring muscle is two joint muscles and is certainly exposed to large length changes. The hamstring constitutes three large muscles that are semi-tendinosis, semi-membranous and biceps femoris. They are positioned in the posterior compartment of the thigh and act on the hip and knee joint as hip extensors and knee flexors. Flexibility dysfunction is a common problem encountered by general as well as athletic population specifically in hamstring.

The tightness of hamstring muscle not only causes decrease range of motion but it can also be a reason for many musculoskeletal dysfunctions. Tightness results in adaptive shortening of the contractile and non-contractile elements of the muscle. The two-joint muscles are more prone to shortening. The tightness of hamstring affects the lumbo-pelvic rhythm. Moreover the tight hamstring restricts the anterior tilting of pelvic in the position of spinal flexion which causes increase tension of muscles and ligaments in the lumbar area resulting in aggravated compressive load on lumbar spine. It also has an indirect effect on sacroiliac joint stability causing Sacro Iliac Joint pain.

The most common method of treatment is to initially feel for areas of soft tissue injury. Then, the tissue is taken from a shortened position to fully lengthened position with a specific hand contact on the soft tissue. This allows the contact to pass longitudinally along the soft tissue fibers and the lesion. The goal is to break up adhesions that may have formed from scarring within the soft tissue. In addition, ART also aims to restore soft tissue structures that feel strained or inflexible to their original healthy condition. The use of ART is becoming a commonality in the restoration of soft tissue injuries, especially in the world of competitive sports.

Active release technique therapy for the hamstrings is intended to relieve pain and lessen tightness and support the hamstring to reappear in its normal condition.

Mulligan's bent leg raise (BLR) is a stretching technique which is a modern progression in the treatment of hamstring tightness. It is indicated in hamstring tightness patients with backache having restricted or painful straight leg raise (SLR), leg pain above knee and it is very beneficial in the patients having gross bilateral limitations of straight leg raise. It stretches the lower extremity muscles in combination of hamstring, adductors and rotators. The BLR technique consists of three repetitions of pain-free isometric contraction of the hamstrings, performed in five progressively greater positions of hip flexion.

ELIGIBILITY:
Inclusion Criteria:

* Patients having Low Back Pain due to hamstring tightness.
* Patients having Sacro Iliac Joint pain due to hamstring tightness.
* 20-40-degree active knee extension loss with hip in 90-degree flexion

Exclusion Criteria:

* Fractures of hip and knee.
* Patients with hamstring injury in past 2 years.
* Hypermobility of lower limb joint.
* Neurological abnormalities.
* Tumors
* Infection
* Medical history of injury to back
* Inflammatory conditions (rheumatoid arthritis, ankylosing spondylitis)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test | four weeks
  The Active Knee Extension test is used to measure the length of hamstring, with normal values of knee motion to within 20֯degree of full extension being quoted. The patient lies in supine position on a plinth and flexes his knee and hip to 90֯. The therapist monitors the position of the femur with his hand. The patient was asked to extend his involved leg as far as possible; keeping his foot relaxed, and holds the position for 5sec. The angle of knee extension was measured using a standard goniometer
Lower extremity functional scale | four weeks
  The Lower extremity functional scale is a questionnaire consisting of 20 questions, used to assess a person's ability to perform everyday tasks. The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.
Visual Analogue Scale (VAS). | four weeks
  This tool is used to measure the intensity of pain. The patient marks the intensity of pain on scale ranging 0 to 10. Where 0 is no pain and 10 describes worst ever type of pain
Modified sit and reach test | four weeks
  This test is used to assess the flexibility of hamstring and lower back. For the Modified Sit and Reach, the participants will be seated on the floor with head, back and hip against a wall (90◦ angle at hip joint), with both legs fully extended and the feet placed against the box. In this position, the participant will be required to place hand over hand and reach out level with the measurement scale, keeping the head, back, and hips in contact with the wall, with only scapular abduction performed. Then the finger to-box distance will be measured as the distance between the fingertips and the point at which the feet rested against the box (point 35 of the scale).

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Aziz Bhatti Shaheed Hospital, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No